CLINICAL TRIAL: NCT06629909
Title: Safety and Feasibility of Human Umbilical Cord Mesenchymal Stem Cell-Derived Secretome in the Treatment of Liver Cirrhosis: a Comprehensive Evaluation of Fibrosis Reduction, Immunomodulation, and Hepatic Regeneration a Single Center, Non-randomized, Phase I Clinical Trial
Brief Title: Safety and Feasibility of Human Umbilical Cord Mesenchymal Stem Cell-Derived Secretome in the Treatment of Liver Cirrhosis: a Comprehensive Evaluation of Fibrosis Reduction, Immunomodulation, and Hepatic Regeneration: a Single Center, Randomized, Phase I Clinical Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baermed (Other)
Collaborators: Tarumanagara University (Other); Liver Clinic Prof Ali Sulaiman (Unknown); Pelni Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-UTHREC/UNTAR/VIII/2024
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; secretome; stem cells; HUCMSC
MeSH Terms: conditions — Liver Cirrhosis | interventions — Secretome; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Secretome Injection (Experimental): patient will receive secretome injection every two weeks for four months
  Interventions: Drug: Secretome
- Best Treatment Practice (No Intervention): patient will receive hepatoprotector drugs and Urodeoxycolate acid for four months

INTERVENTIONS:
Drug: Secretome — 3 ml Injection of secretome for 8 times two weeks apart
  Other Names: hepatoprotector drugs; ursodeoxycholic acid
  Arms: Secretome Injection

SUMMARY:
The goal of this clinical trial is to learn if Human Umbilical Cord Mesenchymal Stem Cell (HUCMSC) derived secretome injection is safe and effective in patient with liver cirrhosis. The main questions it ams to answer are:

1. How safe is secretome Injection as an adjuvant therapy for liver cirrhosis patients?
2. How effective is secretome injection in liver fibrosis 6 months after injection?
3. Does secretome injection improve liver function after 6 months after Injection?
4. Does secretome injection affect Child Turcotte Pugh score?
5. How does secretome affect pro inflammatory and anti Inflammatory cytokine in patient with liver cirrhosis?
6. How does secretome injection affect the quality of life in live cirrhosis patient?
7. What is the relationship between secretome injection and encephalopathy? Researchers will compare secretome injection group (patients who recieve secretome injections) to best practice treatment group (patient who receive supportive treatment including hepatoprotector and ursodeoxycolic acid)

Researchers will compare the intervention group (patients who are injected with HUCMSC derived secretome) and control group (patients who are only monitored and given their usual drugs)

Patients will:

Be injected with secretome or take hepatoprotector and ursodeoxycolic acid every 2 weeks for 4 months. Do several test such us fibroscan, stroop test, psychometric hepatic encephalopathy score, short form 36 questionnaire, IL-6, TNF alfa and blood test for albumin, SGOT, SGPT, direct bilirubin, indirect bilirubin, INR, creatinine, ureum, hemoglobin, hematocrite, leukocyte, and thrombocyte.

Visit the clinic once every two weeks to receive drugs and treatment for 4 months.

Follow up visit to review treatment progress on 3rd months (2 weeks post treatment), 7th months (3 months post treatment),10th months (6 months post treatment)

ELIGIBILITY:
Inclusion Criteria:

* Age above 17 years, both men and women
* Patient is willing to participate and sign informed consent
* Patient is diagnosed with liver cirrhosis confirmed by clinical examination and diagnostic imaging
* Liver cirrhosis patient with Child-Pugh Class B
* Patient is in a stable condition without life threatening complications such as active gastrointestinal bleeding, severe infection, severe renal failure (eGFR&amp>30) at time of registration
* Patient is not receiving experimental drugs for liver cirrhosis for the past 6 months
* Patient is able and willing to comply with research protocol including follow up visits and evaluations

Exclusion Criteria:

* Patient with uncontrolled psychiatric disorders
* Patient who is diagnosed with hepatic or non- hepatic malignancy
* Lactating and pregnant patient
* Patient who has allergy or hypersensitivity reaction towards secretome

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Fibroscan and M2BPGi six month after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Patients achieved a response if there are changes in Fibroscan and M2BPGi after secretome injections within six months.best outcome when the M2BPGi Fibroscan decrease, worst outcome when the M2BPGi and Fibroscan increase
Changes in Complete Blood Count and Kidney function after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Secretome is safe If hemoglobin and hematocrit, leukocyte, platelet, ureum, and creatinine are still in normal level after secretome injection (best outcome)
  Secretome is not safe if hemoglobin and hematocrit, leukocyte, platelet, ureum, and creatinine are out of the normal level after secretome injection (worst outcome)
Changes of albumin, SGOT and SGPT levels in six month after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Patients achieved a response if there are changes in albumin, SGOT and SGPT levels after secretome injections within six months.best outcome when the albumin, SGOT and SGPT decrease, worst outcome when the albumin, SGOT and SGPT increase

SECONDARY OUTCOMES:
Changes of CTP and MELD score in six month after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Patients achieved a response if there are changes in CTP and MELD score after secretome injections within six months.best outcome when the CTP and MELD score decrease, worst outcome when the CTP and MELD score increase
Changes of IL-6 and TNF-α levels in six month after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Patients achieved a response if there are changes in IL-6 and TNF-α levels after secretome injections within six months.best outcome when the IL-6 and TNF-α decrease, worst outcome when the IL-6 and TNF-α increase
Changes of Stroop test dan PHES score in six month after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Patients achieved a response if there are changes inStroop test dan PHES score after secretome injections within six months.best outcome when the Stroop test dan PHES score increase, worst outcome when the Stroop test dan PHES score decrease
Changes of SF-36 questionnaire score in six month after secretome injections | From enrollment to the end of treatment at 4 months, From enrollment to the end of study at 10 months
  Patients achieved a response if there are changes in SF-36 questionnaire score after secretome injections within six months.best outcome when the SF-36 questionnaire score increase, worst outcome when the SF-36 questionnaire score decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Clinic Prof Ali Sulaiman, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Case Report Form (all collected IPD)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication with no end date

REFERENCES:
- See also: Related Info — https://stemcellres.biomedcentral.com/articles/10.1186/s13287-017-0752-6
- See also: Related Info — http://link.springer.com/10.1007/978-3-319-99328-7_2
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fncel.2020.590960/full
- See also: Related Info — https://bioscmed.com/index.php/bsm/article/view/80
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26647219/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35464407
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32883343/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6006340/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6429346/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9575787/
- See also: Related Info — https://bmcgastroenterol.biomedcentral.com/articles/10.1186/s12876-017-0618-5
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38219719/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35285104/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36359492/
- See also: Related Info — https://www.nature.com/articles/s41598-017-14358-0
- See also: Related Info — https://stemcellres.biomedcentral.com/articles/10.1186/s13287-015-0072-7
- See also: Related Info — http://stemcellres.biomedcentral.com/articles/10.1186/s13287-017-0635-x
- See also: Related Info — https://stemcellres.biomedcentral.com/articles/10.1186/s13287-021-02284-y
- See also: Related Info — https://stemcellres.biomedcentral.com/articles/10.1186/s13287-022-03109-2
- See also: Related Info — https://www.degruyter.com/document/doi/10.1515/revneuro-2017-0069/html
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/37383529
- See also: Related Info — https://www.oaepublish.com/articles/jca.2023.15
- See also: Related Info — https://link.springer.com/10.1007/s11033-021-06360-7
- See also: Related Info — https://stemcellres.biomedcentral.com/articles/10.1186/s13287-020-01891-5
- See also: Related Info — http://www.biomed.cas.cz/physiolres/pdf/2019/68_S131.pdf
- See also: Related Info — https://www.nature.com/articles/srep27791
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fcell.2022.1005926/full
- See also: Related Info — https://www.eurekaselect.com/191031/article
- See also: Related Info — http://www.spandidos-publications.com/10.3892/ijmm.2021.4848
- See also: Related Info — https://doi.org/10.21203/rs.3.rs-293044/v1
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22320928
- See also: Related Info — https://doi.org/10.3389/fimmu.2022.833878
- See also: Related Info — https://doi.org/10.3389/fimmu.2022.880523
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34948088